CLINICAL TRIAL: NCT01833442
Title: Randomized Controlled Meditation Trial for Treating OCD Comparing Kundalini Yoga Meditation Versus the Relaxation Response
Brief Title: Randomized Controlled Meditation Trial for Treating OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Euripedes C. Miguel, Chairmain of psychiatry Departament of University os Sao Paulo, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Ipq0704/10br
Record Dates: First submitted 2012-12-04; First posted 2013-04-16 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: OCD
Keywords: OCD; YBOCS

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kundalini Yoga Meditation (Active Comparator): Kundalini Yoga Meditation is going to be use as therapy for OCD, and it will be compare with Relaxation Response Meditation.
  Interventions: Behavioral: Kundalini Yoga Meditation
- Relaxation Response Meditation (Active Comparator): Relaxation Response Meditation is going to be use as therapy for OCD, and it will be compare with Kundalini Yoga Meditation.
  Interventions: Behavioral: Relaxation Response Meditation

INTERVENTIONS:
Behavioral: Kundalini Yoga Meditation — The trial will compare two very different meditation protocols. After the 4.5 month the patients will be reevaluated, and all patients will be merged together into a single group. Patients will then receive 9 - 12 more months of the meditation protocol.
  Arms: Kundalini Yoga Meditation
Behavioral: Relaxation Response Meditation — The trial will compare two very different meditation protocols. After the 4.5 month the patients will be reevaluated, and all patients will be merged together into a single group. Patients will then receive 9 - 12 more months of the meditation protocol.
  Arms: Relaxation Response Meditation

SUMMARY:
The trial objective is to compare two very different meditation protocols (Kundalini Yoga and Relaxation Response meditation techniques) to help the OCD treatment.

DETAILED DESCRIPTION:
The proposed trial comparing the two different meditation protocols is expected to have two phases: 0-month to 4.5-month period where we compare the Kundalini Yoga protocol with Relaxation Response meditation technique, both on the primary efficacy variable using the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) and some if not most of the secondary variables using The Dimensional Yale-Brown Obsessive Compulsive Scale (DY-BOCS), Clinical Global Impressions (CGI), Profile of Mood States (POMS), Beck Anxiety Inventory (Beck-A), Beck Depression Inventory (Beck-D), and SF-36 Health Status Questionnaire (SF36). Participants will go to the hospital once a week for a 1,5 hour meditation class.After 4.5-months, all patients will be evaluated and merged together into a single group. Patients will then receive 09 to 12 more months of the meditation protocol. The investigators are expecting to recruit 50 to 60 patients to start. Patients will be blinded to the content of the protocol in the other group at baseline and until one group shows greater efficacy on the primary efficacy variable. The intake physician will be blinded to the treatment groups of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of OCD for at least 6 months.
* A minimum score of 16 on the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) for the 10-item total score at the baseline screening will be required.
* The patient must sign and been provided with a copy of an Assent Form for their reference.

Exclusion Criteria:

* Psychoactive prescription medications other than those prescribed for OCD.
* Spinal problems, or other physically limiting problems.
* Clinical diagnosis of hypertension, or other cardiovascular problems.
* Clinical diagnosis of Parkinson's disease.
* Clinical diagnosis of major depressive disorder with psychotic features, schizophrenia, bipolar disorder, mental retardation, anorexia nervosa, bulimia nervosa, autistic disorder, Asperger's disorder and other forms of pervasive developmental disorder, or traumatic brain.
* Clinical diagnosis of Tourette's Syndrome.
* Patients without regular and reliable transportation to the study site.
* Patients who choose not to participate in meditation and/or chanting (out loud or silently) for personal or religious reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The Yale-Brown Obsessive Compulsive Scale (YBOCS) | Up to 16 months
  The Yale-Brown Obsessive Compulsive Scale, sometimes referred to as Y-BOCS, is a test to rate the severity of obsessive-compulsive disorder (OCD) symptoms.

SECONDARY OUTCOMES:
The Dimensional Yale-Brown Obsessive-Compulsive Scale (DY-BOCS) | Up to 16 months
  The Dimensional Yale-Brown Obsessive-Compulsive Scale (DY-BOCS): an instrument for assessing obsessive-compulsive symptom dimensions.
Clinical Global Impressions (CGI) | Up to 16 months
Profile of Mood States (POMS) | Up to 16 months
Beck Anxiety Inventory (Beck-A) | Up to 16 months
Beck Depression Inventory (Beck-D) | Up to 16 months
SF-36 Health Status Questionnaire (SF36) | Up to 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Euripedes C Miguel, PHD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Shannahoff-Khalsa D, Fernandes RY, Pereira CAB, March JS, Leckman JF, Golshan S, Vieira MSR, Polanczyk GV, Miguel EC, Shavitt RG. Kundalini Yoga Meditation Versus the Relaxation Response Meditation for Treating Adults With Obsessive-Compulsive Disorder: A Randomized Clinical Trial. Front Psychiatry. 2019 Nov 11;10:793. doi: 10.3389/fpsyt.2019.00793. eCollection 2019. PMID 31780963